CLINICAL TRIAL: NCT01196429
Title: A Phase II Evaluation of Temsirolimus (CCI-779) (NCI Supplied Agent: NSC# 683864,) in Combination With Carboplatin and Paclitaxel Followed by Temsirolimus Consolidation as First-Line Therapy in the Treatment of Clear Cell Carcinoma of the Ovary
Brief Title: Temsirolimus, Carboplatin, and Paclitaxel as First-Line Therapy in Treating Patients With Newly Diagnosed Stage III-IV Clear Cell Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02653; NCI-2011-02653 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000684262; GOG-0268; GOG-0268 (Other: NRG Oncology); GOG-0268 (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2010-09-04; First posted 2010-09-08 (Estimated); Results first posted 2017-05-03 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Ovarian Clear Cell Cystadenocarcinoma; Stage III Ovarian Cancer; Stage IV Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Carboplatin; Docetaxel; Paclitaxel; Taxes; temsirolimus; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (paclitaxel, carboplatin, temsirolimus, docetaxel) (Experimental): Patients receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1 and temsirolimus IV on days 1 and 8. Treatment repeats every 3 weeks for 6 courses. Patients then receive consolidation therapy comprising temsirolimus IV on days 1, 8, and 15. Treatment repeats every 3 weeks for 11 courses in the absence of disease progression or unacceptable toxicity.
  NOTE: * For circumstances in which docetaxel should be substituted for paclitaxel, docetaxel is given IV over 1 hour.
  Interventions: Drug: Carboplatin; Drug: Docetaxel; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Drug: Temsirolimus

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplat; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Docetaxel — Given IV
  Other Names: RP56976; Taxotere; Taxotere Injection Concentrate
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Drug: Temsirolimus — Given IV
  Other Names: CCI-779; CCI-779 Rapamycin Analog; Cell Cycle Inhibitor 779; Rapamycin Analog; Rapamycin Analog CCI-779; Torisel

SUMMARY:
This phase II trial studies how well temsirolimus, carboplatin, and paclitaxel as first-line therapy works in treating patients with newly diagnosed stage III-IV clear cell ovarian cancer. Temsirolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as carboplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving temsirolimus with combination chemotherapy may be an effective treatment for ovarian cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the activity of the study regimen as measured by the proportion of patients who are alive and progression-free for at least 12 months after study entry in patients with newly diagnosed stage III or IV clear cell ovarian cancer in the following populations: patients in the United States (U.S.) and worldwide (outside of Japan) and patients in Japan.

II. To compare progression-free survival in newly diagnosed stage III or IV clear cell ovarian cancer patients in patients in the U.S. and worldwide (outside of Japan) versus patients in Japan.

SECONDARY OBJECTIVES:

I. To characterize the duration of overall survival and progression-free survival in each population.

II. To examine the frequency and severity of adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 4 in each population.

III. To estimate the rate of objective tumor response in patients with measurable disease.

TERTIARY OBJECTIVES:

I. To explore whether immunohistochemical (IHC) expression of components of the mammalian target of rapamycin (mTOR) signaling pathway (phosphatase and tensin homolog [PTEN], total and phosphorylated protein kinase B [Akt], as well as, ATP-binding cassette, sub-family C [CFTR/MRP], member 3 [ABCC3] [MRP3], ATPase, H+ transporting, lysosomal accessory protein 1 [AB CF2], cyclin E, and vascular endothelial growth factor [VEGF]) are associated with outcome, nationality or clinical characteristics.

II. To explore whether there is any differences in differential gene expression profiles between U.S. and worldwide (outside of Japan) versus Japanese patients.

OUTLINE:

Patients receive paclitaxel* intravenously (IV) over 3 hours and carboplatin IV over 30 minutes on day 1 and temsirolimus IV on days 1 and 8. Treatment repeats every 3 weeks for 6 courses. Patients then receive consolidation therapy comprising temsirolimus IV on days 1, 8, and 15. Treatment repeats every 3 weeks for 11 courses in the absence of disease progression or unacceptable toxicity.

NOTE: * For circumstances in which docetaxel should be substituted for paclitaxel, docetaxel is given IV over 1 hour.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have stage III or IV clear cell ovarian cancer; primary tumors must be at least 50% clear cell histomorphology in order to be eligible; in addition, the tumors should be negative for expression of Wilms tumor 1 (WT-1) antigen and estrogen receptor (ER) antigen by immunohistochemistry; appropriate tissue sections to confirm stage and histologic classification of cell type must be sent to Gynecologic Oncology Group (GOG) for central pathology review; immunohistochemical stained slides for ER and WT-1 antigen must be also be submitted to GOG for pathology review
* Patients who have met the pre-entry requirements
* Patients must have signed an approved informed consent and authorization permitting release of personal health information
* Patients with a GOG performance status of 0, 1, or 2
* Patients must be entered between 2 and 12 weeks after initial surgery; performed for the combined purpose of diagnosis, staging and cytoreduction
* Patients should be free of active infection requiring antibiotics (with the exception of uncomplicated urinary tract infection [UTI])
* Absolute neutrophil count >= 1,500/mcl
* Platelets >= 100,000/mcl
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) =< 2.5 times institutional upper limit of normal (< 5 times upper limit of normal [ULN] for subjects with liver metastases)
* Alkaline phosphatase =< 2.5 times institutional upper limit of normal (< 5 times ULN for subjects with liver metastases)
* Creatinine =< 1.5 x institutional upper limit of normal, grade 1 per CTCAE v. 4.0
* Cholesterol =< 350 mg/dL (fasting)
* Triglycerides =< 400 mg/dL (fasting)
* Albumin >= 3.0 g/dL
* Prothrombin time (PT) such that international normalized ratio (INR) is =< 1.5 (or an in-range INR, usually between 2 and 3, if a patient is on a stable dose of therapeutic warfarin for management of venous thrombosis including pulmonary thrombo-embolus)
* Partial thromboplastin time (PTT) < 1.2 times the upper limit of normal
* Neurologic function (sensory and motor) =< CTCAE grade 1

Exclusion Criteria:

* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer, are excluded if there is any evidence of other malignancy being present within the last five years; patients are also excluded if their previous cancer treatment contraindicates this protocol therapy
* Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis are excluded; prior radiation for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than five years prior to registration, and the patient remains free of recurrent or metastatic disease
* Patients who have received prior chemotherapy for any abdominal or pelvic tumor including neo-adjuvant chemotherapy for their clear cell ovarian cancer
* Patients with primary peritoneal and fallopian tube carcinoma are not eligible
* Previous treatment with an mTOR inhibitor (sirolimus, temsirolimus, everolimus), paclitaxel, or carboplatin
* Patients cannot be receiving enzyme-inducing antiepileptic drugs (enzyme-inducing antiepileptic drugs [EIAEDs]; e.g., phenytoin, carbamazepine, phenobarbital) nor any other cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) inducer such as rifampin or St. John's Wort; use of agents that potently inhibit CYP3A4 (and hence may raise temsirolimus levels), such as ketoconazole, is discouraged, but not specifically prohibited; the appropriateness of use of such agents is left to physician discretion; strong CYP3A4 inhibitors are prohibited
* Patients receiving any investigational agents
* Patients with severely impaired lung function defined as a diffusion lung capacity for carbon monoxide (DLCO) =< 50% of the normal predicted value and/or oxygen (O2) saturation =< 88% at rest on room air
* Patients with symptomatic congestive heart failure of New York Heart Association class III or IV, unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction =< 6 months of start of study drug, serious uncontrolled cardiac arrhythmia or any other clinically significant disease
* Patients with active bleeding or pathologic conditions that carry high risk of bleeding, such as known bleeding disorder, coagulopathy, or tumor involving major vessels
* Patients on maintenance corticosteroids are ineligible with the exception of short term use (fewer than 5 days)
* Patients with baseline requirement for oxygen
* Patients with serious concomitant illness which, in the opinion of the treating physician, will place patient at unreasonable risk from therapy on this protocol
* Patients who are pregnant or nursing; patients of childbearing potential must agree to use contraceptive measures during study therapy and for at least six months after completion of study therapies
* Patients with poorly controlled diabetes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2010-08; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Farley, Principal Investigator — NRG Oncology
Locations (145):
- United States (121):
  - Saint Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Florida Hospital Orlando, Orlando, Florida
  - Memorial University Medical Center, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Sudarshan K Sharma MD Limted-Gynecologic Oncology, Hinsdale, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Cadence Cancer Center in Warrenville, Warrenville, Illinois
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Saint Vincent Oncology Center, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium CCOP, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa Oncology Research Association CCOP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Walter Reed Army Medical Center-Olney, Olney, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium CCOP, Ann Arbor, Michigan
  - Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Gynecologic Oncology of West Michigan PLLC, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Michiana Hematology Oncology PC-Niles, Niles, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Lakeland Hospital, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Mercy Hospital-Joplin, Joplin, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Winthrop University Hospital, Mineola, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Tulsa Cancer Institute, Tulsa, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - M D Anderson Cancer Center CCOP Research Base, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - PeaceHealth Medical Group PC, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Skagit Valley Hospital Regional Cancer Care Center, Mount Vernon, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Group Health Cooperative-Seattle, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Northwest Hospital, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Olympic Medical Cancer Care Center, Sequim, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Rockwood Cancer Treatment Center-DHEC-Downtown, Spokane, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
- Japan (17):
  - Tohoku University School of Medicine, Sendai, Aoba-ku
  - Kure National Hospital, Kure, Hiroshima
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Hyogo Cancer Center, Akashi, Hyōgo
  - Iwate Medical University School of Medicine, Morioka, Iwate
  - Kagoshima City Hospital, Kagoshima, Kagoshima-ken
  - Niigata University Medical and Dental Hospital, Niigata, Niigata
  - University of the Ryukyus Hospital-Col Health Scnc, Nakagami-gun, Okinawa
  - Shizuoka Cancer Center, Shizuoka, Suntou
  - Keio University, Shinjuku-ku, Tokyo
  - Shikoku Cancer Center, Matsuyama
  - National Kyushu Cancer Center, Minamiku
  - Jikei University School of Medicine, Minato-ku, Tokyo
  - Kinki University, Osaka, Osaka
  - Saitama Medical University International Medical Center, Saitama
  - National Cancer Center Hospital, Tokyo
  - Tottori University, Tottori
- South Korea (7):
  - Keimyung University-Dongsan Medical Center, Jung-Ku, Daegu
  - National Cancer Center-Korea, Goyang-si, Gyeonggi-do
  - Samsung Medical Center, Seoul, Korea
  - Seoul National University Hospital, Seoul
  - Gangnam Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Korea Cancer Center Hospital, Seoul

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on 8/30/2010 and closed to accrual on 1/6/2014.
Pre-assignment Details: Additional details about the interventions administered were not included because these are groups (not arms).
Groups:
- US/Korea; Japan: Temsirolimus (CCI-779) 25mg IV Days 1 and 8, Carboplatin AUC= 6 IV Day 1 and Paclitaxel 175 mg/m2 IV on Day 1 every 3 weeks for cycles 1-6 or disease progression. Followed by consolidation therapy with temsirolimus (CCI-779) 25 mg weekly on Days 1, 8 and 15 every 3 weeks cycles 7-17 or until disease progression
Period: Overall Study
Arm/Group | US/Korea | Japan
Started | 45 | 45
Completed | 42 | 45
Not Completed | 3 | 0
Not completed — Ineligible - inadequate pathology | 1 | 0
Not completed — Ineligible - wrong cell type | 1 | 0
Not completed — Refused - Never Treated | 1 | 0

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients
Groups:
- Total: Total of all reporting groups
Arm/Group | US/Korea | Japan | Total
Number analyzed (Participants) | 42 | 45 | 87
Age, Customized [Number; unit: participants]
  20-29 years | 1 | 1 | 2
  30-39 years | 2 | 3 | 5
  40-49 years | 12 | 9 | 21
  50-59 years | 21 | 21 | 42
  60-69 years | 6 | 8 | 14
  70-79 years | 0 | 3 | 3
  80-89 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 45 | 87
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Who Are Alive and Progression-free for at Least 12 Months After Study Entry in Patients With Newly Diagnosed Stage III or IV Clear Cell Ovarian Cancer in the Following Populations: Patients in the U.S./Worldwide and Japan
Description: Progression of target lesions (TL) was a >=20% increase in the sum of the diameters of TL, taking as reference the smallest sum on study (including the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must demonstrate an absolute increase >=5 mm. Progression of non-target lesions (NTL) as defined as appearance of >=1 new lesions or unequivocal progression of existing NTL. Unequivocal progression should not normally trump target lesion status; it must be representative of overall disease status change, not a single lesion increase. Clear progression of only NTL is exceptional, but the opinion of the treating physician should prevail in such circumstances, and the progression status should be later confirmed by a review panel (or Principal Investigator). Progression of TL, unequivocal progression of NTL, or new lesions constitutes progression. This description is abbreviated; see the RECIST 1.1 manuscript for further details.
Time Frame: Tumor scans were done every other cycle for the first 6 months; then every 3 months x2; then every 6 months thereafter; and at any other time if clinically indicated or signs suggestive of progressive disease or rising levels; for up to 5 years.
Population: Eligible and Treated Patients
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- US/Korea; Japan: Progression-free survival (PFS) was defined as the period from study entry until disease progression, death, or the last date of contact. Patients censored prior to 12 months were considered failures in this analysis. Progression was based on RECIST 1.1
Arm/Group | US/Korea | Japan
Number analyzed (Participants) | 42 | 45
percentage of participants | 43 [31 to 55] | 53 [41 to 65]

2. Primary Outcome: Compare Progression-free Survival in Newly Diagnosed Stage III or IV Clear Cell Ovarian Cancer Patients in Patients in the U.S. and Worldwide (Outside of Japan) Versus Patients in Japan.
Description: Progression-free survival (PFS) was defined s the period from study entry until disease progression, death, or the last date of contact. Progression was based on Response Evaluation Criteria In Solid Tumors (RECIST) 1.1. Outcome measure data not reported because protocol stated "If the combination is declared active (i.e. HO is rejected) in one or both of the populations, the two populations will be compared with respect to PFS using a logrank test stratified by optimal/suboptimal disease status." The combination was not declared active in either population.
Time Frame: Tumor scans were done every other cycle for the first 6 months;then every 3 mnths x2;then every 6 mnths thereafter; and at any other time if clinically indicated based on symptoms or physical signs suggesting progressive dx or rising serum tumor marker le
Population: The protocol stated "if the combination is declared active (i.e., HO is rejected) in one or both of the populations, the two populations will be compared with respect to PFS using a logrank test stratified by optimal/suboptimal disease status". The combination was not declared active in either population.
Arm/Group | US/Korea | Japan
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Frequency and Severity of Toxicity
Description: Grade 3 or higher adverse events were graded by CTC AE v4
Time Frame: Each cycle while on treatment
Population: Eligible and Treated Patients
Measure: Number; unit: participants
Arm/Group | US/Korea | Japan
Number analyzed (Participants) | 42 | 45
participants
  Neutrophil count decreased | 36 | 42
  White blood cell decreased | 27 | 32
  Anemia | 9 | 13
  Platelet count decreased | 10 | 10
  Hypertension | 4 | 10
  hypertriglyceridemia | 6 | 7
  Mucositis oral | 5 | 5
  Febrile neutropenia | 4 | 5
  Diarrhea | 6 | 2
  Hypokalemia | 3 | 4
  Hyperglycemia | 4 | 2
  Abdominal pain | 3 | 1
  Lymphocyte count decreased | 2 | 2
  Nausea | 1 | 2
  Urinary tract infection | 3 | 0
  GGT increased | 0 | 3
  Edema limbs | 2 | 0
  Fatigue | 1 | 1
  Fever | 1 | 1
  Non-cardiac chest pain | 2 | 0
  Cholesterol high | 0 | 2
  Weight gain | 2 | 0
  Hypoalbuminemia | 1 | 1
  Hyponatremia | 2 | 0
  Hypophosphatemia | 0 | 2
  Peripheral Sensory neuropathy | 0 | 2
  Cough | 2 | 0
  Dyspnea | 2 | 0
  Pharyngeal mucositis | 0 | 2
  Rash maculo-papular | 1 | 1
  Colonic perforation | 0 | 1
  Constipation | 1 | 0
  Ileus | 1 | 0
  Oral pain | 1 | 0
  Small intestinal obstruction | 1 | 0
  Vomiting | 1 | 0
  Pain | 1 | 0
  Cholecystitis | 1 | 0
  Hepatobiliary disorders-other | 0 | 1
  Appendicitis perforated | 0 | 1
  Kidney infection | 1 | 0
  Lung infection | 1 | 0
  Peripherl nerve infection | 1 | 0
  Pharyngitis | 0 | 1
  Skin infection | 1 | 0
  Infections and infestations -other | 1 | 0
  Alanine aminotransferase increased | 0 | 1
  Aspartate aminotransferase increased | 0 | 1
  Creatiine increased | 0 | 1
  Anorexia | 0 | 1
  Dehydration | 1 | 0
  Hypermagnesemia | 0 | 1
  Back Pain | 1 | 0
  Bone Pain | 1 | 0
  Flank pain | 1 | 0
  Pain in Extremity | 1 | 0
  Dizziness | 0 | 1
  Paresthesia | 1 | 0
  Vasovagal reaction | 1 | 0
  Anxiety | 1 | 0
  Dysparenuia | 1 | 0
  Pneumonitis | 0 | 1
  Sore throat | 1 | 0
  Hypotension | 1 | 0
  Lymphocele | 1 | 0

4. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) was defined as the period from study entry until disease progression, death, or the last date of contact. Progression was based on RECIST 1.1
Time Frame: Tumor scans were done every other cycle for the first 6 months; then every 3 months x 2; then every 6 mths thereafter; and at any other time if clinically indicated based on symptoms or physical signs suggestive of progressive disease or rising tumor mark
Population: Eligible and Treated Patients
Measure: Median (90% Confidence Interval); unit: months
Groups:
- US/Korea: Patients enrolled from the U.S.and Korea
- Japan: Patients enrolled from Japan
Arm/Group | US/Korea | Japan
Number analyzed (Participants) | 42 | 45
months | 11.0 [6.1 to 14.3] | 12.1 [9.5 to 16.6]

5. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the duration of time from study entry to time of death or the date of last contact.
Time Frame: Every cycle during treatment, then every 3 months for the first 2 years, then every six months for the next three years and then annually for the next 5 years.
Population: Eligible and Treated Patients
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | US/Korea | Japan
Number analyzed (Participants) | 42 | 45
months | 22.6 [19.2 to 36.3] | 25.6 [21.4 to NA] — Not reached, but is >37.1 months.

6. Secondary Outcome: Objective Tumor Response
Description: Complete and Partial Tumor Response by RECIST 1.1. RECIST1.1 is a multi-page paper, and response is defined in the protocol across multiple pages, so it is not practical to define response here.
Time Frame: Every other cycle for first 6 months; then every 3 months for two years; then every six months for the next three years; and at any other time if clinically indicated based on symptoms or physical signs suggestive of progressive disease or rising serum tu
Population: Eligible and Treated Patients
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | US/Korea | Japan
Number analyzed (Participants) | 42 | 45
percentage of participants | 54 [32 to 74] | 71 [51 to 85]

ADVERSE EVENTS:
Time Frame: Study Treatment
Arm/Group | US/Korea | Japan
Serious Adverse Events (participants affected / at risk) | 11/42 | 8/45
Other Adverse Events (participants affected / at risk) | 42/42 | 45/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | US/Korea (N=42) | Japan (N=45)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 2 | 0
Mucositis Oral (Gastrointestinal disorders) | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 1 | 0
Fever (General disorders) | 1 | 1
Hepatobiliary Disorders - Other (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 2 | 0
Kidney Infection (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0
Appendicitis Perforated (Infections and infestations) | 0 | 1
Platelet Count Decreased (Investigations) | 0 | 2
Neutrophil Count Decreased (Investigations) | 5 | 1
White Blood Cell Decreased (Investigations) | 1 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 | 0
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal Mucositis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | US/Korea (N=42) | Japan (N=45)
Lymph Node Pain (Blood and lymphatic system disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 42 | 45
Febrile Neutropenia (Blood and lymphatic system disorders) | 3 | 5
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 3 | 4
Sinus Tachycardia (Cardiac disorders) | 3 | 3
Chest Pain - Cardiac (Cardiac disorders) | 0 | 3
Vertigo (Ear and labyrinth disorders) | 0 | 2
Tinnitus (Ear and labyrinth disorders) | 9 | 0
Hearing Impaired (Ear and labyrinth disorders) | 2 | 0
Ear Pain (Ear and labyrinth disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Hypoparathyroidism (Endocrine disorders) | 1 | 0
Watering Eyes (Eye disorders) | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 7
Blurred Vision (Eye disorders) | 8 | 0
Dry Eye (Eye disorders) | 2 | 2
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 7 | 0
Dyspepsia (Gastrointestinal disorders) | 8 | 1
Colonic Perforation (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 19 | 21
Diarrhea (Gastrointestinal disorders) | 24 | 26
Cheilitis (Gastrointestinal disorders) | 0 | 3
Vomiting (Gastrointestinal disorders) | 16 | 18
Bloating (Gastrointestinal disorders) | 4 | 0
Stomach Pain (Gastrointestinal disorders) | 0 | 8
Anal Mucositis (Gastrointestinal disorders) | 2 | 2
Rectal Mucositis (Gastrointestinal disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 17 | 8
Rectal Hemorrhage (Gastrointestinal disorders) | 2 | 0
Oral Dysesthesia (Gastrointestinal disorders) | 1 | 0
Mucositis Oral (Gastrointestinal disorders) | 25 | 40
Gastrointestinal Disorders - Other (Gastrointestinal disorders) | 2 | 0
Anal Pain (Gastrointestinal disorders) | 0 | 1
Oral Hemorrhage (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 5
Gastrointestinal Pain (Gastrointestinal disorders) | 1 | 1
Gingival Pain (Gastrointestinal disorders) | 1 | 0
Oral Pain (Gastrointestinal disorders) | 4 | 0
Abdominal Distension (Gastrointestinal disorders) | 4 | 0
Nausea (Gastrointestinal disorders) | 28 | 26
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 2 | 1
Rectal Pain (Gastrointestinal disorders) | 1 | 0
Hemorrhoidal Hemorrhage (Gastrointestinal disorders) | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 2 | 2
Ascites (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 3
Esophageal Pain (Gastrointestinal disorders) | 0 | 1
Dental Caries (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 3
General Disorders And Administration Site Conditio (General disorders) | 1 | 0
Pain (General disorders) | 10 | 3
Malaise (General disorders) | 2 | 24
Localized Edema (General disorders) | 1 | 0
Injection Site Reaction (General disorders) | 1 | 1
Infusion Site Extravasation (General disorders) | 0 | 6
Flu Like Symptoms (General disorders) | 4 | 14
Edema Trunk (General disorders) | 1 | 1
Non-Cardiac Chest Pain (General disorders) | 4 | 0
Edema Limbs (General disorders) | 12 | 22
Facial Pain (General disorders) | 1 | 0
Edema Face (General disorders) | 4 | 7
Fatigue (General disorders) | 36 | 19
Fever (General disorders) | 8 | 8
Gait Disturbance (General disorders) | 1 | 0
Chills (General disorders) | 7 | 1
Infusion Related Reaction (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Allergic Reaction (Immune system disorders) | 3 | 3
Infections And Infestations - Other (Infections and infestations) | 3 | 0
Upper Respiratory Infection (Infections and infestations) | 4 | 5
Vulval Infection (Infections and infestations) | 0 | 1
Skin Infection (Infections and infestations) | 3 | 4
Sinusitis (Infections and infestations) | 3 | 0
Rash Pustular (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 3
Peripheral Nerve Infection (Infections and infestations) | 1 | 0
Otitis Media (Infections and infestations) | 1 | 0
Papulopustular Rash (Infections and infestations) | 0 | 1
Nail Infection (Infections and infestations) | 2 | 0
Mucosal Infection (Infections and infestations) | 2 | 0
Lung Infection (Infections and infestations) | 2 | 1
Paronychia (Infections and infestations) | 0 | 8
Eye Infection (Infections and infestations) | 1 | 1
Small Intestine Infection (Infections and infestations) | 1 | 0
Gum Infection (Infections and infestations) | 0 | 2
Vaginal Infection (Infections and infestations) | 2 | 0
Urinary Tract Infection (Infections and infestations) | 6 | 2
Bladder Infection (Infections and infestations) | 0 | 5
Lip Infection (Infections and infestations) | 1 | 1
Wound Dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 2
Wound Complication (Injury, poisoning and procedural complications) | 0 | 1
Bruising (Injury, poisoning and procedural complications) | 2 | 2
Weight Loss (Investigations) | 8 | 14
Weight Gain (Investigations) | 10 | 10
Serum Amylase Increased (Investigations) | 0 | 1
Platelet Count Decreased (Investigations) | 39 | 41
Lymphocyte Count Decreased (Investigations) | 5 | 2
Inr Increased (Investigations) | 0 | 2
Ggt Increased (Investigations) | 0 | 9
Creatinine Increased (Investigations) | 2 | 7
Cholesterol High (Investigations) | 22 | 30
Neutrophil Count Decreased (Investigations) | 42 | 44
Cpk Increased (Investigations) | 0 | 2
Blood Bilirubin Increased (Investigations) | 1 | 1
White Blood Cell Decreased (Investigations) | 42 | 45
Aspartate Aminotransferase Increased (Investigations) | 10 | 16
Alkaline Phosphatase Increased (Investigations) | 11 | 11
Alanine Aminotransferase Increased (Investigations) | 12 | 13
Activated Partial Thromboplastin Time Prolonged (Investigations) | 0 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 5 | 3
Hyponatremia (Metabolism and nutrition disorders) | 9 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 16 | 2
Hypokalemia (Metabolism and nutrition disorders) | 18 | 5
Hypoglycemia (Metabolism and nutrition disorders) | 3 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 8 | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 9 | 8
Hypertriglyceridemia (Metabolism and nutrition disorders) | 23 | 31
Hypernatremia (Metabolism and nutrition disorders) | 3 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 3
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 19 | 22
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 7 | 1
Anorexia (Metabolism and nutrition disorders) | 20 | 30
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 13 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 12 | 27
Muscle Weakness Upper Limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 2 | 0
Joint Range Of Motion Decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 4 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 6 | 0
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 5 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 6 | 7
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 | 25
Musculoskeletal And Connective Tissue Disorder - (Musculoskeletal and connective tissue disorders) | 1 | 2
Neoplasms Benign, Malignant And Unspecified (Incl (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Vasovagal Reaction (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 2 | 0
Somnolence (Nervous system disorders) | 0 | 3
Presyncope (Nervous system disorders) | 1 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 28 | 43
Peripheral Motor Neuropathy (Nervous system disorders) | 3 | 5
Paresthesia (Nervous system disorders) | 6 | 1
Neuralgia (Nervous system disorders) | 2 | 2
Memory Impairment (Nervous system disorders) | 2 | 0
Movements Involuntary (Nervous system disorders) | 1 | 0
Hypersomnia (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 15 | 10
Dysgeusia (Nervous system disorders) | 5 | 24
Sinus Pain (Nervous system disorders) | 1 | 0
Dysesthesia (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 7 | 2
Cognitive Disturbance (Nervous system disorders) | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0
Personality Change (Psychiatric disorders) | 1 | 0
Restlessness (Psychiatric disorders) | 2 | 0
Libido Decreased (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 13 | 11
Depression (Psychiatric disorders) | 9 | 2
Confusion (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 14 | 0
Anorgasmia (Psychiatric disorders) | 1 | 0
Urinary Urgency (Renal and urinary disorders) | 1 | 0
Urinary Incontinence (Renal and urinary disorders) | 2 | 0
Urinary Tract Pain (Renal and urinary disorders) | 7 | 0
Urinary Frequency (Renal and urinary disorders) | 7 | 1
Renal Calculi (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 2 | 4
Hematuria (Renal and urinary disorders) | 1 | 1
Cystitis Noninfective (Renal and urinary disorders) | 0 | 3
Chronic Kidney Disease (Renal and urinary disorders) | 1 | 0
Vaginal Pain (Reproductive system and breast disorders) | 1 | 0
Vaginal Hemorrhage (Reproductive system and breast disorders) | 2 | 1
Pelvic Pain (Reproductive system and breast disorders) | 1 | 0
Vaginal Discharge (Reproductive system and breast disorders) | 1 | 0
Vaginal Inflammation (Reproductive system and breast disorders) | 1 | 0
Dyspareunia (Reproductive system and breast disorders) | 4 | 0
Respiratory, Thoracic And Mediastinal Disorders - (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Voice Alteration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus Disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 9
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pharyngeal Mucositis (Respiratory, thoracic and mediastinal disorders) | 0 | 8
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal Mucositis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Laryngeal Inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 15
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 14 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 5
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Skin And Subcutaneous Tissue Disorders - Other (Skin and subcutaneous tissue disorders) | 2 | 5
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 9
Skin Ulceration (Skin and subcutaneous tissue disorders) | 4 | 0
Skin Induration (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 1
Skin Atrophy (Skin and subcutaneous tissue disorders) | 0 | 1
Rash Acneiform (Skin and subcutaneous tissue disorders) | 14 | 18
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 12
Periorbital Edema (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar-Plantar Erythrodysesthesia Syndrome (Skin and subcutaneous tissue disorders) | 0 | 4
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 14 | 18
Skin Hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Nail Ridging (Skin and subcutaneous tissue disorders) | 2 | 4
Nail Loss (Skin and subcutaneous tissue disorders) | 0 | 4
Nail Discoloration (Skin and subcutaneous tissue disorders) | 3 | 5
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 4 | 6
Bullous Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 30 | 39
Vasculitis (Vascular disorders) | 0 | 5
Thromboembolic Event (Vascular disorders) | 1 | 0
Lymphocele (Vascular disorders) | 1 | 0
Lymphedema (Vascular disorders) | 5 | 7
Hypotension (Vascular disorders) | 2 | 2
Hypertension (Vascular disorders) | 15 | 25
Hot Flashes (Vascular disorders) | 9 | 4
Hematoma (Vascular disorders) | 0 | 1
Flushing (Vascular disorders) | 1 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less